CLINICAL TRIAL: NCT03857178
Title: A Multi-country Study on the Prescription Patterns of Short Acting Beta-2 Agonist (SABA) and Its Potential Effects on Asthma Control: A Cross-Sectional Study on SABA Use in Asthma
Brief Title: SABINA INTERNATIONAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589SR00002
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The aim of the study is to describe the prescribing pattern of the different types of medications which are used to treat asthma, across multiple countries.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥12 years-old
2. Documented diagnosis with Asthma as per medical records.
3. Have had ≥3 consultations with the HCP at study start date
4. After full explanation, a patient or legal guardian must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Patient with a diagnosis of chronic obstructive pulmonary disease or other chronic respiratory disease different from Asthma.
2. An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The selection of sites and investigators will be made with the aim to achieve representativeness in the way asthma is managed in each participating country. The study will include patients from either primary care centres, or specialist centres involved in the management of asthma, or a mix of both within a country to ensure representativeness.
Sampling Method: Non-Probability Sample
Enrollment: 8617 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
The main outcome will be a categorisation of SABA prescription in asthma patients. | 12 months retrospective from index date
  Mild asthma patients will be categorised into 5 groups according to the number of SABA and ICS prescriptions in the 12 months prior to their index date (initial exposure window):
  1. No prescriptions for asthma inhalers
  2. Appropriate SABA prescription with no ICS
  3. Appropriate SABA prescription with ICS
  4. SABA over-prescription with no ICS
  5. SABA over-prescription with ICS
  Moderate/severe asthma patients will be categorised into 2 groups according to the number of SABA and ICS prescriptions in the 12 months prior to their index date:
  1. Appropriate SABA prescription on top of maintenance therapy
  2. SABA over-prescription on top of maintenance therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, San Salvador, Argentina

REFERENCES:
- [Derived] Tan DHY, Tan TL, Tan WH, Choong C, Beekman MJHI, Khor JH, Kumar SS, Wong GR, Lim HF. SABA prescriptions and asthma management practices in Singapore: results from a cross-sectional, observational SABINA III study. BMJ Open. 2024 Jun 10;14(6):e064245. doi: 10.1136/bmjopen-2022-064245. PMID 38858145
- [Derived] Alzaabi A, Al Busaidi N, Pradhan R, Shandy F, Ibrahim N, Ashtar M, Khudadah K, Hegazy K, Samir M, Negm M, Farouk H, Al Khalidi A, Beekman M. Over-prescription of short-acting beta2-agonists and asthma management in the Gulf region: a multicountry observational study. Asthma Res Pract. 2022 Jul 7;8(1):3. doi: 10.1186/s40733-022-00085-5. PMID 35799290
- [Derived] Bateman ED, Price DB, Wang HC, Khattab A, Schonffeldt P, Catanzariti A, van der Valk RJP, Beekman MJHI. Short-acting beta2-agonist prescriptions are associated with poor clinical outcomes of asthma: the multi-country, cross-sectional SABINA III study. Eur Respir J. 2022 May 5;59(5):2101402. doi: 10.1183/13993003.01402-2021. Print 2022 May. PMID 34561293
- See also: This is the CSR of the study. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589SR00002&attachmentIdentifier=b42e4dc0-e8ac-4e40-b05c-4ef8cf69a41d&fileName=CSR_SABINA_V_0.6_CTT_with_Milestones_Combined.pdf&versionIdentifier=